CLINICAL TRIAL: NCT06379555
Title: Wrist Fractures Management With Arthroscopic Assistance Under Walant - Exploratory Study
Acronym: WALANPOIGNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02756-39
Record Dates: First submitted 2024-04-17; First posted 2024-04-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Wrist Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walanpoigne (Experimental): This arm will combine WALANT anesthesia WALANT with arthroscopy to reduce a joint fracture of the wrist
  Interventions: Procedure: Walanpoigne

INTERVENTIONS:
Procedure: Walanpoigne — Intervention will combine WALANT anesthesia with arthroscopy to reduce a joint fracture of the wrist

SUMMARY:
Wrist articular fractures are more difficult to treat and rehabilitation takes longer. Furthermore, these joint fractures are frequently accompanied by ligament lesions of the carpal bones.

For these reasons, it is strongly recommended to check the interior of the wrist joint. This check can be done with wrist arthroscopy. Therefore, fracture reduction can be improved, "step of stairs" can be eliminated under arthroscopic control and ligament rupture of carpal bones can be treated.

WALANT anesthesia (Wide Awake Local Anesthesia No Tourniquet) designates a new local anesthesia technique. This technique which allows to maintain the arm or fingers mobility offers several significant advantages:

* Greater precision of the surgical procedure.
* A reduction in discomfort, risks and related adverse effects to anesthesia.
* Faster recovery.

WALANT technique is very comfortable for patient and fits perfectly with principles of Enhanced Recovery in Surgery.

In this context, this study is based on the hypothesis that it is possible to combine arthroscopy and the WALANT anesthesia technique for reducing wrist fractures

DETAILED DESCRIPTION:
Wrist fractures are common. Most often, when speaking about wrist fracture, this means distal radius fracture, the radius being one of the two forearm bones and most often affected in cases of fracture. A fracture is articular when the fracture line "goes down" in the joint.

These fractures are more difficult to treat and rehabilitation takes longer because it is necessary to ensure that joint surface is perfectly reduced, this means that there are no "stair steps" in the joint. Furthermore, these joint fractures are frequently accompanied by ligament lesions of the carpal bones.

For all these reasons, it is strongly recommended to check the interior of the wrist joint. This check can be done with wrist arthroscopy. Arthroscopy not only allows for a complete assessment of lesions but also to treat most of them. Therefore, fracture reduction can be improved, "step of stairs" can be eliminated under arthroscopic control and a ligament rupture of carpal bones can be treated.

WALANT anesthesia (Wide Awake Local Anesthesia No Tourniquet) designates a new local anesthesia technique which is based on administration, in association with local anesthetic (lidocaine), of a medicine (epinephrine) which limits bleeding and allows to dispense with a tourniquet. The local anesthetic administration allows to maintain the arm or fingers mobility, while having complete anesthesia. This technique offers several significant advantages:

* Greater precision of the surgical procedure. In fact, bleeding limitation and the patient's state of cooperation allow a greater surgical precision.
* A reduction in discomfort, risks and related adverse effects to anesthesia.
* Faster recovery.

WALANT technique is very comfortable for patient and fits perfectly with principles of Enhanced Recovery in Surgery. Several studies have shown that it is possible to reduce distal radius fractures under WALANT anesthesia. As for wrist arthroscopy, this is a classic technique for controlling inside of the wrist joint, allowing not only to have an overall view of wrist injuries but also to treat most of them.

In this context, this study is based on the hypothesis that it is possible to combine arthroscopy and the WALANT anesthesia technique for reducing wrist fractures

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 and < 70 years
* Patient with a displaced articular fracture of the distal radius (unilateral wrist fracture)
* Patient treated on ambulatory way
* Patient affiliated to or beneficiary of a social security system
* French speaking patient, having signed informed consent

Exclusion Criteria:

* Patient with previous infection or wrist bone surgery
* Patient with multiple fractures or with bilateral wrist fractures
* Patient with associated fracture with the wrist fracture
* Patient with "pathological" bone
* Protected patient: adult under guardianship, curatorship or other protection legal, deprived of liberty by judicial or administrative decision
* Patient hospitalized without consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Failure percentage | Day 1
  A failure is defined by the impossibility of achieving the surgery under WALANT anesthesia. Practically, this translates either to stopping the procedure, either by intra-operative sedation (Protoxide nitrogen, deep hypnosis, general anesthesia) in emergency

SECONDARY OUTCOMES:
Pain assessment | Day 1, 7 and 30
  Pain will be assessed with a VAS (Visual Analogic Scale). Minimum value is 0 and maximum value is 10. 0 means no pain whereas higher scores mean more and more pain.
Patient experience | Day 1
  Patient experience will be evaluated using the e-satis questionnaire. Minimum value is 0 and maximum value is 100. 0 means patient is not satisfied whereas higher scores mean patient is more and more satisfied.
Wrist mobility | Day 7 and 30
  Wrist mobility will be assessed with flexion/extension and pronosupination (measured in degrees with the goniometer)
Functional characteristics of the wrist | Day 7 and 30
  Functional characteristics of the wrist will be assessed with PWRE (Patient-Rated Wrist Evaluation) questionnaire. Each question is rated from 0 to 10. Higher scores mean a worse outcome.
Functional characteristics of the wrist | Day 7 and 30
  Functional characteristics of the wrist will be assessed with QuickDash questionnaire. Each question is rated from 1 to 5. Higher scores mean a worse outcome.
Complications | Day 1 to Day 30
  Complications will be assessed with collection of adverse events, particularly intraoperative bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Les Franciscaines (Hôpital privé de Versailles), Versailles, France

IPD SHARING:
Plan to Share IPD: No